CLINICAL TRIAL: NCT03608293
Title: Particulate Air Pollution : Smoker Extracellular Vesicles Influence on Human Bronchial Epithelial Cells
Brief Title: Smoker Extracellular Vesicles Influence on Human Bronchial Epithelial Cells
Acronym: Aerotox-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC-P0014
Record Dates: First submitted 2018-07-24; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Smokers; Human Bronchial Epithelial Cells; Lung Pathogenesis; Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers (Experimental): Smokers outpatients at the Pneumology service from the HôpitalSaint-Philibert (Lomme, France) to whom a bronchoalveolar lavage will be performed
  Interventions: Diagnostic Test: Broncho Alveolar Lavages (BAL)
- Non smokers (Active Comparator): Non smokers outpatients at the Pneumology service from the HôpitalSaint-Philibert (Lomme, France) to whom a bronchoalveolar lavage will be performed
  Interventions: Diagnostic Test: Broncho Alveolar Lavages (BAL)

INTERVENTIONS:
Diagnostic Test: Broncho Alveolar Lavages (BAL) — BEAS-2 B cells are exposed to EVs isolated from BAL of smokers and non-smokers.

SUMMARY:
Cigarette smoking is a habit that has spread all over the world and is a significant risk factor for many diseases including cardiovascular disease, chronic obstructive pulmonary disease(COPD),asthma and lung cancer.

Evaluation and understanding of tobacco health effects are of major interest worldwide and answer to important societal concerns.

Identification of new biomarkers of exposure to tobacco smoke potentially implicated in COPD or lung carcinogenesis would allow a better observation of tobacco exposed population, thanks to screening establishment at reversible stages of pathological processes.

In this study, we question whether cigarettes smoking alters miRNA profiles of extracellular vesicles (EVs) present in human broncho alveolar lavages (BALs), which could affect surrounding normal bronchial epithelial cells status.

DETAILED DESCRIPTION:
Extracellular vesicles (EVs) include a variety of nanoscale membranous vesicles (exosomes, microvesicles, microparticles). EVs are released into the interstitial fluid from a wide variety of normal or diseased cells.

Analysis of EVs and their content maybe useful as disease biomarkers as they reflect the contents of cells of origin, differ between normal and diseased tissue and can be reliably detected.

EVs may thus act as biomarkers of diverse pathologies like cancer, and detection of these biomarkers maybe applied to early diagnosis or assessment of prognosis in patients with cancer. EVs indeed contain both mRNAs and non-coding RNAs, such as small regulatory microRNAs (miRNAs).

ELIGIBILITY:
Inclusion Criteria:

* >18 year-old

Exclusion Criteria:

* Lack of informed consent
* Drug treatment
* Professional exposure
* Evolutive pregnancy
* Bradycardia
* Respiratory assistance required,
* Diagnosed respiratory distress (e.g. COPD, asthma)
* Infectious pneumopathy
* Bronchial cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Quantification of target mRNA expression in human bronchial epithelial cells (BEAS-2 B) exposed to EVs isolated from LBA of patients | Through the study completion, an average of 48 months
  Quantitative polymerase chain reaction (RT-qPCR) for determination of mRNA expression

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Gosset, MD, Principal Investigator — GHICL